CLINICAL TRIAL: NCT00725647
Title: A Study of the Value of Plasma N-terminal proBNP Concentrations for Diagnosing Patent Ductus Arteriosus in Preterm Babies.
Brief Title: Plasma N-terminal proBNP Concentrations and Patent Ductus Arteriosus in Preterm Babies
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: National Health Service, United Kingdom (Other Government); Medical Research Council (Other Government)
Responsible Party: Dr Santhanakrishnan Ramakrishnan (Principal investigator), St George's Healthcare NHS Trust
Other Study IDs: 04/Q0803/98
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Ductus Arteriosus, Patent
Keywords: N terminal B type natriuretic peptide; echocardiography; diagnosis; atrial natriuretic peptides; preterm infant
MeSH Terms: conditions — Ductus Arteriosus, Patent; Disease; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated PDA: Infants who had a PDA which the attending physicians treated medically or surgically.

SUMMARY:
Premature babies are affected by a condition known as "patent ductus arteriosus" in which the ductus arteriosus (a normal structure) fails to close after birth as it should. A very large ductus can put extra strain on the heart and lungs, making the baby's breathing dependent on a mechanical ventilator. Attending physicians can close the duct with medical\or surgical treatment but assessing whether this is justified can be difficult. The physician usually bases this decision on assessment of the baby's general condition and an ultrasound evaluation of the heart (called an "echocardiogram") but the last is particularly dependent on availability of skilled operators.

The investigators have examined whether blood levels of a hormone called B-type natriuretic peptide (Nt pro-BNP)in the first week of life predict the need to treat a ductus arteriosus. This hormone is produced by the heart if it is under strain. If the test is helpful it could reduce dependence of physicians on echocardiography by skilled operators.

Babies who were recruited had blood samples collected on days 1, 2, 3 and 7 for measurement of Nt pro-BNP. Each baby also had an echocardiogram performed between the fifth and seventh day of life. Decisions about treatment of the duct were made by attending physicians independent of the study. Physicians, investigators and echocardiographers were blinded to knowledge of the Nt pro-BNP concentration. Nt pro-BNP was also measured before and after treatment in all babies who had a PDA treated and echocardiography performed to confirm closure.

Receiver operating characteristics (ROC) curves were used to assess the predictive value of Nt pro-BNP for samples collected at each time point. The investigators also compared the Nt pro-BNP levels in samples collected before and after treatment to assess the usefulness of Nt pr-BNP as an indicator of duct closure.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies under 34-weeks gestation admitted to the neonatal intensive care unit

Exclusion Criteria:

* Known structural heart abnormality other than PDA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants in a tertiary level neonatal intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santhanakrishnan Ramakrishnan, MB MRCPCH, Principal Investigator — St George's Healthcare NHS Trust; Anthony F Williams, MB FRCPCH, Study Director — St George's, University of London

REFERENCES:
- [Result] Ramakrishnan S, Heung YM, Round J, Morris TP, Collinson P, Williams AF. Early N-terminal pro-brain natriuretic peptide measurements predict clinically significant ductus arteriosus in preterm infants. Acta Paediatr. 2009 Aug;98(8):1254-9. doi: 10.1111/j.1651-2227.2009.01315.x. Epub 2009 Apr 30. PMID 19432837